CLINICAL TRIAL: NCT01963481
Title: Phase II Trial of Exemestane With Immunomodulatory Cyclophosphamide in ER and/or PR-positive and HER2/Neu Negative Metastatic Breast Cancer
Brief Title: Exemestane and Cyclophosphamide for Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-00761
Record Dates: First submitted 2013-10-11; First posted 2013-10-16 (Estimated); Results first posted 2020-03-17 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Metastatic Beast Cancer
Keywords: hormonal therapy; immunotherapy
MeSH Terms: interventions — exemestane; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Exemestane and cyclophosphamide (Experimental): A treatment cycle is defined as 4 weeks:
  One tablet (25 mg) of exemestane and one tablet (50 mg) of cyclophosphamide given daily by mouth until disease progression or unacceptable adverse events.
  Interventions: Drug: Exemestane; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Exemestane
  Other Names: Aromasin
Drug: Cyclophosphamide
  Other Names: Cytoxan; CTX

SUMMARY:
This phase II trial studies how well exemestane and cyclophosphamide work in treating patients with estrogen receptor (ER) -positive, progesterone receptor (PR) -positive, and human epidermal growth factor receptor (HER)2-negative stage IV breast cancer.

DETAILED DESCRIPTION:
Estrogen can cause the growth of breast cancer cells. Hormone therapy using exemestane may fight breast cancer by blocking the use of estrogen by the tumor cells. Low dose cyclophosphamide may also stimulate the white blood cells, including natural killer cells, for instance by decreasing the suppressor (regulatory) T-cells. Giving exemestane with cyclophosphamide may be an effective treatment for estrogen receptor-positive, progesterone receptor-positive, and HER2-negative stage IV breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed breast cancer that is ER positive and/or PR positive, and HER2/neu negative and have disease that is metastatic (stage IV)

  * HER2/neu negative disease determined using commercially available/approved assay in local institutional or reference laboratory, according to American Society of Clinical Oncology (ASCO)/College of American Pathologists (CAP) guidelines (IHC 0-1+ or 2+ with HER2/17 ratio on FISH <= 1.8).
  * ER/PR expression performed by standard immunohistochemical assay and classified as ER and/or PR-positive according to ASCO/CAP guidelines (1-100% expression)
  * Histologic and/or cytologic confirmation of metastatic disease is encouraged whenever feasible, furthermore, if feasible, the biopsy should confirm that the metastatic tumor is ER and/or PR positive and HER2/neu negative. For patients in whom histologic biopsy confirmation and/or assessment of ER/PR/HER2 of metastatic disease is not feasible, it is required that the primary tumor be ER and/or PR-positive and HER2/neu negative.
* Measurable disease (RECIST 1.1) or non-measurable (assessable) disease
* Patients must have had progressive disease during at least one line of endocrine therapy for metastatic disease or have recurrent disease while or within 12 months of receiving adjuvant endocrine therapy. Prior treatments accepted include a non-steroidal aromatase inhibitor, tamoxifen, fulvestrant or combinations.
* Patients taking bisphosphonates for bone disease are permitted to enter the trial, but their bone lesions are not considered to be assessable for response, although they are assessable for progression.
* Female or male subjects age >= 18 years.
* Eastern Cooperative Oncology Group (ECOG) performance status 0, 1, or 2.
* Patients must have normal organ and marrow function as defined below:
* absolute neutrophil count >= 1,200/mcL
* platelets >= 100,000/mcL
* hemoglobin >= 9g/dl
* total bilirubin <= 2 X upper limit of normal (ULN) [unless due to Gilbert's disease]
* AST(SGOT) <= 2.5 X ULN
* ALT(SGPT) <= 2.5 X ULN
* creatinine <= 1.5 X ULN
* Patients must be able to swallow and tolerate oral medications.
* Postmenopausal status, defined as 60 years and older, being 45 years and older and having amenorrhea x 12 months or follicle stimulating hormone levels within postmenopausal range, OR having undergone a bilateral oophorectomy.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients may not be receiving any other investigational agents.
* Prior treatment for breast cancer with a steroidal aromatase inhibitor; with the exception of patients who were started on the combination of exemestane with everolimus less than 4 weeks prior to study entry and discontinued everolimus due to poor tolerability.
* Presence of life threatening metastatic visceral disease (defined as extensive hepatic involvement or symptomatic pulmonary lymphangitic spread) or uncontrolled brain metastases.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2013-09; Primary Completion 2017-10-01 (Actual); Study Completion 2017-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sylvia Adams, MD, Principal Investigator — NYU Perlmutter Cancer Center
Locations (1):
- NYU Cancer Center, New York, New York, United States

REFERENCES:
- [Derived] Kwa M, Li X, Novik Y, Oratz R, Jhaveri K, Wu J, Gu P, Meyers M, Muggia F, Speyer J, Iwano A, Bonakdar M, Kozhaya L, Tavukcuoglu E, Budan B, Raad R, Goldberg JD, Unutmaz D, Adams S. Serial immunological parameters in a phase II trial of exemestane and low-dose oral cyclophosphamide in advanced hormone receptor-positive breast cancer. Breast Cancer Res Treat. 2018 Feb;168(1):57-67. doi: 10.1007/s10549-017-4570-4. Epub 2017 Nov 9. PMID 29124456

RESULTS

PARTICIPANT FLOW:
Groups:
- Exemestane and Cyclophosphamide: A treatment cycle is defined as 4 weeks:
  One tablet (25 mg) of exemestane and one tablet (50 mg) of cyclophosphamide given daily by mouth until disease progression or unacceptable adverse events.
  Exemestane
  Cyclophosphamide
Period: Overall Study
Arm/Group | Exemestane and Cyclophosphamide
Started | 23
Completed | 23
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Exemestane and Cyclophosphamide
Number analyzed (Participants) | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 23
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 23
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 23

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) Rate at 3 Months
Description: PFS is defined as the time from first treatment day until objective disease progression or death from any cause. Assessment of disease progression based on Response Evaluation Criteria in Solid Tumor (RESIST) guideline version 1.1 is performed every 12 weeks on study. The percent of participants with PFS at 3 months will be reported.
Time Frame: 3 months
Measure: Number (95% Confidence Interval); unit: percent of participants
Arm/Group | Exemestane and Cyclophosphamide
Number analyzed (Participants) | 23
percent of participants | 50.1 [33.0 to 76.0]

2. Secondary Outcome: Response Rate (RR) - Complete Response and Partial Response
Description: Complete response (CR) is defined as the disappearance of all target lesions, while partial response (PR) is when at least a 30% decrease in the sum of the diameters of target lesions. Evaluation of response is based on RESIST guideline version 1.1. RR is reported as percentage of participants with a CR and/or PR at 2 years.
Time Frame: 2 years
Measure: Number (95% Confidence Interval); unit: percent of participants
Arm/Group | Exemestane and Cyclophosphamide
Number analyzed (Participants) | 23
percent of participants | 26.1 [10.2 to 48.4]

3. Secondary Outcome: Clinical Benefit Rate Score
Description: Clinical benefit rate is defined as the percentage of patients who have achieved objective response or stable disease for at least 24 weeks. Evaluation of response and disease progression is based on RESIST guideline version 1.1. Response and progression are assessed every 12 weeks.
Time Frame: 3 years
Measure: Number (95% Confidence Interval); unit: percent of participants
Arm/Group | Exemestane and Cyclophosphamide
Number analyzed (Participants) | 23
percent of participants | 47.8 [26.8 to 69.4]

ADVERSE EVENTS:
Time Frame: 13.7 Months
Arm/Group | Exemestane and Cyclophosphamide
All-Cause Mortality (participants affected / at risk) | 10/23
Serious Adverse Events (participants affected / at risk) | 10/23
Other Adverse Events (participants affected / at risk) | 0/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Exemestane and Cyclophosphamide (N=23)
pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 10 (23)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-09-12): https://cdn.clinicaltrials.gov/large-docs/81/NCT01963481/Prot_SAP_000.pdf